CLINICAL TRIAL: NCT02295904
Title: Video Analysis of Vaginal Deliveries to Evaluate the Impact of the Support of the Perineum
Brief Title: Video Analysis of Vaginal Deliveries
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.2014-0414
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Birth Trauma
Keywords: perineum; videoanalysis
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Video documentation of vaginal deliveries to evaluate the impact of the support of the perineum

DETAILED DESCRIPTION:
Documentation of support of perineum via video camera, documentation of birth trauma after delivery, record of fetal and maternal parameters as weight, hight, fetal presentation, etc.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women,
* at least 18 years of age (yoa),
* term deliveries (at least 37+0 weeks of gestation),
* vaginal delivery,
* fetal vertex presentation,
* single pregnancy

Exclusion Criteria:

* younger than 18 yoa,
* preterm deliveries,
* cesarean sections,
* fetal malformations,
* maternal disease in form of collagenosis,
* multiples pregnancy,
* vaginal/vulvar/perineal pre-operations (excluding birth trauma),
* perineal birth trauma grade III+IV

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
adequate support of perineum | 12 months
  documentation of support of perineum via video camera during delivery, documentation of birth trauma after delivery, documentation of fetal and maternal parameters as weight, hight, fetal presentation, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kimmich, MD, Principal Investigator — University Hospital Zurich, Division of Obstetrics
Locations (1):
- University Hospital Zurich, Division of Obstetrics, Zurich, Canton of Zurich, Switzerland